CLINICAL TRIAL: NCT04659239
Title: A Randomized, Double-Blinded, Placebo Controlled Phase III Clinical Trial of SARS-CoV-2 Vaccine, Inactivated (Vero Cell) in Adults Aged 18 Years and Above
Brief Title: The Efficacy, Safety and Immunogenicity Study of Inactivated SARS-CoV-2 Vaccine for Preventing Against COVID-19
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Qihan Li, Professor, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 20200404
Record Dates: First submitted 2020-12-05; First posted 2020-12-09 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — SARS-CoV-2 inactivated vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigational Vaccine (Experimental): Participants will receive 2 doses of the inactivated SARS-CoV-2 vaccine (Vero cell) according to the immunization schedule of D0, D14.
  Interventions: Biological: Inactivated SARS-CoV-2 Vaccine (Vero cell)
- Placebo (Placebo Comparator): Participants will receive 2 doses of the placebo according to the immunization schedule of D0, D14.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Inactivated SARS-CoV-2 Vaccine (Vero cell) — The inactivated SARS-CoV-2 vaccine (vero cell) was manufactured by IMBCAMS. Each dose of 0.5ml is for per person per time use.
  Arms: Investigational Vaccine
Biological: Placebo — The placebo was manufactured by IMBCAMS. Each dose of 0.5ml is for per person per time use.
  Arms: Placebo

SUMMARY:
This is a randomized, double-blinded, placebo controlled phase III clinical trial to evaluate the efficacy, safety and immunogenicity of SARS-CoV-2 Vaccine, Inactivated (Vero Cell) in adults aged 18 years and above after 2-dose schedule.

DETAILED DESCRIPTION:
The trial includes two parts, namely the efficacy study and immunogenicity bridging study. A total of 34020 participants will be enrolled, i.e. 32820 for efficacy cohort, and 1200 for domestic immunogenicity cohort in China.

Efficacy study: Participants will be randomly inoculated with two doses of investigational vaccine or placebo according to 1:1 ratio following Day 0-Day 14 immunization schedule and will be observed from the first dose of investigational vaccine to collect symptomatic and laboratory-confirmed COVID-19 cases for the evaluation of the efficacy of the investigational vaccine.

Immunogenicity bridging study: Before inoculating the first dose, 14 days, 6 months and 12 months after the whole-course immunization, blood samples will be taken for determination of neutralizing antibody and IgG antibody against SARS-CoV-2 (ELISA method); and before inoculating the first dose, 6 months and 12 months after the whole-course immunization, blood samples will be taken for detecting specific T cells with the ELISPOT assay with an aim to evaluate immunogenicity and immune persistence.

Safety observations for all participants will be conducted from the first dose to 28 days after the whole-course immunization, and follow-up of SAEs will also be conducted from the first dose to at least 12 months after the whole-course immunization to evaluate the safety of the investigational vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 years and above (including boundary values), both female and male.
2. Legal identification of the participants shall be provided.
3. Participants shall understand the content in the Informed Consent Form (ICF) and the vaccine for administration, sign the ICF voluntarily and are capable of using thermometers and rulers, and filling in diary cards and contact cards as per the requirements.
4. Subject shall be able to communicate well with investigators, understand and comply with the requirements of this study.
5. Participants with oral temperature ≤ 37.9 ℃.
6. Female participants of childbearing potential (defined as any female who has experienced menarche and who is NOT surgically sterile [i.e., hysterectomy, bilateral tubal ligation, or bilateral oophorectomy] or postmenopausal [defined as amenorrhea at least 12 consecutive months]) must agree to be heterosexually inactive OR consistently use any of the following methods of contraception:

   1. Condoms (male or female)
   2. Diaphragm with spermicide
   3. Cervical cap with spermicide
   4. Intrauterine device
   5. Oral or patch contraceptives
   6. Any country regulatory-approved contraceptive method that is designed to protect against pregnancy
   7. Abstinence, as a form of contraception, is acceptable if in line with the participant's lifestyle (other approaches to abstinence are not acceptable).

Exclusion Criteria:

1. Contraindications to commonly used vaccines;
2. History of allergy to any vaccines or drug;
3. Received any vaccine within 1 month before the first dose of vaccination；
4. Serious diseases required to be excluded, including but not limited to history of diseases in nervous system, cardiovascular system, blood and lymphatic system, immune system, kidney, liver, gastrointestinal tract, respiratory system, metabolism, bones and other systems, and a history of malignant tumors;
5. Before immunizing the first dose of investigational vaccine, those who developed acute disease within 2 weeks, or had symptoms of fever or upper respiratory tract infection within 7 days;
6. Those who have a hereditary bleeding tendency or blood coagulation dysfunction, or a history of thrombosis or hemorrhagic disease；
7. Surgical removal of whole or part of spleen for any reason；
8. Those who have undergone surgery within 3 months before signing the ICF or those who plan to undergo surgery during or within 3 months after completion of the trial (including plastic surgery, dental and oral surgery);
9. Those who donated or lost blood (≥400 mL) in the past 3 months, who received blood transfusion or use of blood products, or who plan blood donation during the trial;
10. Those who received other investigational or unregistered products (drugs, vaccines, biological product or devices) in the past 3 months before signing the ICF, or plan to use them during the study.
11. Those who received immunosuppressant therapy within 6 months before signing the ICF, such as long-term systemic glucocorticoid treatment (with systemic glucocorticoid therapy for more than 2 consecutive weeks within 6 months, such as prednisone or similar drugs), but local administration is permitted (such as ointment, eye drops, inhalants, or nasal spray). The local administration should not exceed the recommended dose in the package insert or have any signs of systemic exposure;
12. Participants cannot meet the criteria through the comprehensive physical examination, mainly including:

    * Abnormal vital signs with clinical significance (awakening heart rate <55 beats/min or >100 beats/min, systolic blood pressure ≥140mmHg or diastolic blood pressure ≥90mmHg);
    * Those who tested positive for type 1 or type 2 human immunodeficiency virus (HIV-1/2) antibody, or SARS-CoV-2 nucleic acid;
13. History of COVID-19;
14. Participants who have a positive pregnancy test, or are breastfeeding, or planning pregnancy, or plan to donate sperm or eggs within 12 months from the screening period to the whole-course immunization;
15. Participants who are considered as inappropriate for the trial by investigators.
16. Suspected or known current alcohol or drug dependency.
17. Investigator site personnel directly related to this study and/or their immediate families; immediate family is defined as a spouse, parent, child, or sibling, whether biological or legally adopted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34020 (Estimated)
Dates: Start 2021-01-28 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
The incidence of COVID-19 cases after two-doses of vaccination | From 14 days after the second dose to 1 year after the second dose.
  The incidence of the symptomatic and laboratory-confirmed COVID-19 cases starting from Day 14 after the second dose.
The incidence of solicited AEs. | 7 days after each dose
  The incidence of solicited AEs at the inoculation site (local) and solicited AEs at the non-inoculation site (systemic) within 7 days after each dose

SECONDARY OUTCOMES:
The incidence of COVID-19 cases after at least one dose of immunization. | From the first dose to 1 year after the second dose.
  The incidence of the symptomatic and laboratory-confirmed COVID-19 cases after at least one dose of immunization.
The Geometric Mean Titer (GMT) of neutralizing antibody | 14 days after the whole-course immunization
  The Geometric Mean Titer (GMT) of neutralizing antibody against SARS-CoV-2 14 days after the whole-course immunization.
The Geometric Mean Titer (GMT) of IgG antibody | 14 days after the whole-course immunization
  The Geometric Mean Titer (GMT) of IgG antibody (ELISA method) against SARS-CoV-2 14 days after the whole-course immunization.
The positive rates of neutralizing antibody | 14 days after the whole-course immunization
  The positive rates of neutralizing antibody against SARS-CoV-2 14 days after the whole-course immunization.
The positive rates of IgG antibody | 14 days after the whole-course immunization
  The positive rates of IgG antibody (ELISA method) against SARS-CoV-2 14 days after the whole-course immunization.
The seroconversion rates of neutralizing antibody | 14 days after the whole-course immunization
  The seroconversion rates of neutralizing antibody against SARS-CoV-2 14 days after the whole-course immunization.
The seroconversion rates of IgG antibody | 14 days after the whole-course immunization
  The seroconversion rates of IgG antibody (ELISA method) against SARS-CoV-2 14 days after the whole-course immunization.
The positive rates of neutralizing antibody | 6 months and 12 months after whole-course immunization.
  The positive rates of neutralizing antibody against SARS-CoV-2 6 months and 12 months after whole-course immunization.
The positive rates of IgG antibody | 6 months and 12 months after whole-course immunization.
  The positive rates of IgG antibody (ELISA method) against SARS-CoV-2 6 months and 12 months after whole-course immunization.
The Geometric Mean Titer (GMT) of neutralizing antibody | 6 months and 12 months after whole-course immunization.
  The Geometric Mean Titer (GMT) of neutralizing antibody against SARS-CoV-2 6 months and 12 months after whole-course immunization.
The Geometric Mean Titer (GMT) of IgG antibody | 6 months and 12 months after whole-course immunization.
  The Geometric Mean Titer (GMT) of IgG antibody (ELISA method) against SARS-CoV-2 6 months and 12 months after whole-course immunization.
Specific T cells with ELISPOT assay | 6 months and 12 months after the whole-course immunization
  Detecting specific T cells with ELISPOT assay 6 months and 12 months after the whole-course immunization
The incidence of AEs | From the first dose to 28 days after whole-course immunization.
  The incidence of AEs from the first dose to 28 days after whole-course immunization
The incidence of SAEs | From the first dose to at least 12 months after whole-course immunization.
  The incidence of SAEs from the first dose to at least 12 months after whole-course immunization.
The occurrence of Antibody Dependent Enhancement (ADE)/ Vaccine Enhanced Disease(VED) | From 14 days after the second dose to 1 year after the second dose.
  The occurrence of Antibody Dependent Enhancement (ADE)/ Vaccine Enhanced Disease(VED) that probably related to the laboratory-confirmed COVID-19 from 14 days after the second dose till the end of trial.

OTHER OUTCOMES:
The surrogate endpoint of immunogenicity | From 14 days after the second dose to 1 year after the second dose.
  The correlation between the efficacy of the vaccine and the levels of neutralizing antibody and IgG antibody against SARS-CoV-2.

CONTACTS AND LOCATIONS:
Overall Officials: Yasmin binti Mohamed Gani, PhD, Principal Investigator — Hospital Sungai Buloh; Adilson JW Cavalcante, PhD, Principal Investigator — CEMEC Pesquisa Clinica
Locations (2):
- CEMEC Pesquisa Clinica, São Bernardo do Campo, São Paulo, Brazil
- Hospital Sungai Buloh, Sungai Buloh, Selangor, Malaysia